CLINICAL TRIAL: NCT00813826
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study Evaluating the Efficacy and Tolerability of Oral SLC022 300 mg TID, a Glial Cell Modulating Agent, Versus Placebo in the Treatment of Post Herpetic Neuralgia
Brief Title: Efficacy and Safety Study of SLC022 in Treating Pain Associated With Post Herpetic Neuralgia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Solace Pharmaceuticals (Industry)
Responsible Party: Kevin Pojasek, Senior Director, Development Programs Leader, Solace Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLC022/201
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Postherpetic Neuralgia
Keywords: PHN; Pain after Shingles
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLC022 (Experimental): 300mg TID
  Interventions: Drug: SLC022; Drug: Placebo
- Placebo (Placebo Comparator): Matching placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLC022 — SLC022 150 mg capsule, 900mg daily dose
  Arms: SLC022
Drug: Placebo — Placebo capsule, TID

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SLC022 in treating pain associated with post-herpetic neuralgia (PHN) in recently diagnosed patients.

DETAILED DESCRIPTION:
This study will enroll subjects with established PHN, a stable pain intensity and that meet all other eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 years or older.
2. A history of cutaneous herpes zoster infection and sustained pain associated with the site of the herpes zoster skin rash for >6 months, after onset of the herpes zoster skin rash.
3. Well established consistent pain during baseline phase.
4. Completed a washout period of 7 days for existing pain medications.
5. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
6. A willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Pregnant or breast feeding.
2. Female subjects who are not surgically sterile (hysterectomy or bilateral tubal ligation), postmenopausal for at least one year, or are not willing to practice adequate methods of contraception if of childbearing potential.
3. Previous neurolytic or neurosurgical therapy for PHN.
4. Treatment with local anesthetic nerve blocks within the last 30 days.
5. Failure of an adequate dose of 3 or more first line drug treatments for PHN-related pain due to efficacy.
6. Any other type of pain which may impair the self assessment of the pain due to PHN.
7. Skin conditions in the affected dermatome that could alter sensation.
8. Participation in other studies within 30 days before the current study begins and/or during study participation.
9. Taking CYP1A2 inhibitors such as fluvoxamine, certain fluoroquinolones (e.g., ciprofloxacin, enoxacin, pefloxacin, etc), mexiletine, and zileuton.
10. History of drug or alcohol abuse during the last 5 years.
11. Creatinine clearance <50 mL/min.
12. History of malignancy other than basal cell carcinoma and carcinoma in situ.
13. History of chronic hepatitis B or C, or human immunodeficiency virus (HIV) infection.
14. Clinically significant hepatic, respiratory, hematological, cardiovascular or neurological disease.
15. Immunocompromised state.
16. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-10 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the change in a subject's mean pain score from the baseline period to the end of the treatment period as measured using the 11-point Numerical Rating Scale. | 7 weeks

SECONDARY OUTCOMES:
Determining the safety and tolerability of SLC022 300 mg TID compared to placebo TID in subjects with PHN by measuring changes in vital signs, ECG, hematology and other laboratory values, and subject-reported adverse events. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Pojasek, PhD, Study Director — Solace Pharmaceuticals Inc.
Locations (19):
- United States (19):
  - Sierra Vista, Arizona
  - Mission Viejo, California
  - Orlando, Florida
  - Plantation, Florida
  - Marietta, Georgia
  - Oak Brook, Illinois
  - Shreveport, Louisiana
  - Brockton, Massachusetts
  - Omaha, Nebraska
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Kettering, Ohio
  - Altoona, Pennsylvania
  - Philadelphia, Pennsylvania
  - West Reading, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Midvale, Utah